CLINICAL TRIAL: NCT05113303
Title: Comparative, Case Control, Mono-center PMCF Study on Manual and Navigated Revision Knee Patients After a Minimum Follow-Up of Two Years
Brief Title: COREV 2.0 PMCF-Study on Manual and Navigated Revision Knee Patients
Acronym: COREV
Status: Completed | Type: Observational
Sponsor: Aesculap AG (Industry)
Collaborators: B.Braun Surgical SA (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-2012
Record Dates: First submitted 2021-10-11; First posted 2021-11-09 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Knee Osteoarthritis; Bone; Deformity, Congenital; Prosthesis Failure; Prosthesis-Related Infections
Keywords: Computer Assisted Surgery; Revision; Total Knee Arthroplasty; Joint Alignment; Observational Study; Forgotten Joint Score
MeSH Terms: conditions — Osteoarthritis, Knee; Congenital Abnormalities; Prosthesis Failure; Prosthesis-Related Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- navigation assisted knee revision surgery
  Interventions: Device: Navigated Revision Total Knee Arthroplasty
- manual procedure
  Interventions: Device: Manual Revision Total Knee Arthroplasty

INTERVENTIONS:
Device: Navigated Revision Total Knee Arthroplasty — Patients in the case group receive a Columbus® Revision knee prosthesis, implanted with computer assisted surgery
  Groups: navigation assisted knee revision surgery
Device: Manual Revision Total Knee Arthroplasty — Patients in the control group will correspond to a historical cohort of patients in which manual jig-assisted knee revision was done.
  Groups: manual procedure

SUMMARY:
The Columbus® Revision endoprosthetic system is bearing the CE-mark. This means that within the scope of this observational study the patient will not be subjected to any additional stressful, study-related medical examinations or treatment measures. The treatment will be carried out exclusively according to medical standards. The study therefore only serves the purpose of observing this standard-compliant treatment and specifically documenting it scientifically.

DETAILED DESCRIPTION:
The study's main purpose is the collection of clinical data on the safety and performance of the Columbus® Revision Knee endoprosthesis

ELIGIBILITY:
Inclusion Criteria:

* Patient underwent navigated revision surgery using the Columbus® Revision knee prosthesis (case group)
* Patient underwent conventional manual revision surgery using another implant system (control group)
* Written informed consent

Exclusion Criteria:

* Pregnancy
* Patient Age at time of revision surgery < 18 years
* Allergy to any prosthesis component

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients in the case group will be recruited consecutively. No selection besides the inclusion and exclusion criteria will take place. The following criteria are applicable for the inclusion of study patients:
  Patients in the control group will correspond to a historical cohort of patients in which manual jig-assisted knee revision was done. A minimum of two years follow up will be necessary to be included.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2024-03-24 (Actual)

PRIMARY OUTCOMES:
Compare the final joint line height between groups after the surgical restoration of native joint line height of revision implants | Comparison of final joint line height before the surgery with height at the 3 months follow-up
  Joint line height will be assessed using the systematic, comparative x-ray analysis

SECONDARY OUTCOMES:
Maintenance of Hip knee Ankle Angle | Comparison of HKA before the surgery with HKA at 3 months and 2 years follow-up
  The HKA within 3 degrees of neutral has been used as the essential outcome measure in TKA.
Forgotten Joint Score | At final follow-up at least 2 years after surgery
  The FJS Knee was designed to assess patient outcome in patients undergoing conservative or operative treatment of the knee. These PRO questionnaires focus on patients' awareness of a specific joint in everyday life. In 12 Items the awareness for the artificial joint is assessed by the patient, each on a five point scale (Never / Almost Never / Seldom / Sometimes / Mostly)
WOMAC Score | At final follow-up at least 2 years after surgery
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is a widely used, proprietary set of standardized questionnaires used by health professionals to evaluate the condition of patients with osteoarthritis of the knee and hip, including pain (5 items), stiffness (2 items), and physical functioning (17 items) of the joints. Each item is assessed by the patient on a five point scale (none / slight / moderate / severe / extreme)
KSS Score | At final follow-up at least 2 years after surgery
  The KSS is an examiner--administrated standard clinical evaluation tool reporting results for patients undergoing TKA. It separates findings in the operated knee (kKSS) score from findings related to the patient's function (fKSS), which might be affected by co-morbidities. The two sub-scores are reported separately ranging from 0 points (worst result) to 100 points (best results), as well as summarized score, total KSS. Final grading of total KSS results Scores of 160 to 200 will be rated as excellent, 140 to 159 as good, 120 to 139 as fair, and less than 120 as poor.
Implant survival | Until final follow-up at least 2 years after surgery
  Survival in the sense of this study is defined as a removal or exchange of any revision implant components including the removal or exchange of the PE meniscus component. Secondary interventions at the index knee e.g. secondary patella replacement do not count as a revision if no further exchange of the former implant components occur.
  The revision-free survival rate is the performance indicator of the product under investigation and confirms the clinical outcome of the knee prosthesis. Information on survival of the implant will be collected until the last follow-up of the study patients took place.
Documentation of Adverse events/serious adverse events | over the whole course of the study from surgery until final follow-up at least 2 years after surgery
  During the course of the study, any upcoming intra- or postoperative (serious) adverse device events or effects related or not related to the product under investigation, will be documented in the dedicated Case Report Forms The total number of AEs will be summarized and further evaluated by the sponsor Recorded complications will be categorized and analyzed in order to assess the safety of the investigational product

OTHER OUTCOMES:
Descriptive analysis of Radiological assessment | from discharge until final follow-up at least 2 years after surgery
  All follow-up imaging exams will be obtained according to the radiographic protocol of the hospital and the set routine. Imaging will be used to evaluate the implant status as well as device condition and potential presence of device-related Adverse Events including fracture, wear, loosening or radiolucencies, as well as the parameters of joint line restoration, rotational alignment and posterior condylar offset.

CONTACTS AND LOCATIONS:
Overall Officials: Emilio Larrazabal Raluy, MD, Principal Investigator — Hospital Universitario Cruces, Spain; Igor Gonzales, MD, Principal Investigator — Hospital Universitario Cruces, Spain
Locations (1):
- Hospital Universitario Cruces, Barakaldo, Bizkaia, Spain